CLINICAL TRIAL: NCT05968443
Title: Observational, Retrospective Clinical Study in Patients Undergoing Ophthalmic Surgery Using Dafilon® Suture Material (Dafilon® USP (United States Pharmacopeia) Sizes From 8/0 to 11/0)
Brief Title: Dafilon® Suture Material in Patients Undergoing Ophthalmic Surgery
Acronym: OPHTHADA
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1913
Record Dates: First submitted 2023-07-17; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Eye Diseases
Keywords: Ophthalmologic Surgery
MeSH Terms: conditions — Eye Diseases | interventions — Ophthalmologic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ophthalmic surgery — any ophthalmic surgery using Dafilon® suture

SUMMARY:
This is an observational, retrospective postmarket clinical follow-up study and includes all patients who underwent any ophthalmic surgery using Dafilon® suture in the selected centres between 2018 and 2020, therefore no sample size can be given but the planned sample size shall be at least 200 eyes (around 100 patients depending on the number of operated eyes per patient) to conduct meaningful subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated between 2018 - 2020 undergoing any ophthalmic surgery using Dafilon® suture material (Dafilon® USP (United States Pharmacopeia) sizes from 8/0 to 11/0) at the participating hospital

Exclusion Criteria:

* No exclusion criteria have been set

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent any ophthalmic surgery using Dafilon® suture in the participating centre between 2018 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Number of Suture material complications | up to the retrospective examination (2 to 4 years postoperatively)
  Suture material complications needing suture removal or reinterventions (Re-suturing due to wound dehiscence)

SECONDARY OUTCOMES:
Number of Intra-operative complications | intraoperatively
  Number of Intra-operative complications as documented in the patient's record
Number of Post-operative complications | up to the retrospective examination (2 to 4 years postoperatively)
  Cumulative number of Post-operative complications including Haemorrhage, inflammation and tissue reaction, corneal lesion, retraction, granuloma, and contracture at the postoperative follow-up examination
Incidence of recurrence | up to the retrospective examination (2 to 4 years postoperatively)
  Cumulative number of recurrencies

CONTACTS AND LOCATIONS:
Overall Officials: Hamidah H Budin, Dr., Principal Investigator — KPJ Tawakkal KL Specialist Hospital
Locations (1):
- KPJ Tawakkal KL Specialist Hospital, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No